CLINICAL TRIAL: NCT00320372
Title: A Long-term, Prospective, Observational, Multi-center Patient Outcome Registry to Collect Data in Patients With Treatment-resistant Depression (TRD) Who Are Currently in a Major Depressive Episode.
Brief Title: Treatment-Resistant Depression Registry
Status: Completed | Type: Observational
Sponsor: Cyberonics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TRD Registry; NCT00657215 (obsolete NCT alias)
Record Dates: First submitted 2006-05-01; First posted 2006-05-03 (Estimated); Results first posted 2015-12-23 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-12

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Treatment-resistant Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1. 500 VNS Patients: VNS Patients - Treatment-resistant depression patients treated with VNS Therapy.
- 2. 300 Non-VNS Patients: Non-VNS Patients - Treatment-resistant depression patients not receiving VNS Therapy.

SUMMARY:
This registry will collect information about patients with treatment-resistant depression (TRD) who are currently in a major depressive episode. For the purposes of this study, TRD is defined as an ongoing depression lasting at least 2 years or that has recurred at least 3 times, to include the current episode, during the patient's lifetime AND has not adequately responded to 4 or more adequate antidepressive treatments. The registry will follow the clinical course and outcomes for patients with TRD who are treated with and without adjunctive (used along with other treatments for depression) vagus nerve stimulation (VNS) therapy.

DETAILED DESCRIPTION:
Enrollment of TRD patients treated with VNS Therapy will consist of patients originally enrolled in the registry as well as patients who have completed the D-21 Dosing Study and are enrolled in the Registry for Long-Term Follow-up. Sites will maintain a screening log of all patients who have been screened for original TRD Registry patients.

Please note that because this is a post-approval registry, Cyberonics does not cover the cost of VNS Therapy implantation.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with a current major depressive episode according to DSM-IV-TR criteria.
* For D-21 patients only who have completed the D-21 dosing Study without any D-21 inclusion and exclusion protocol deviation.
* Patient has been in the current depressive episode for 2 years or longer, or has had at least 3 lifetime episodes including the current MDE.
* Patient has had an inadequate response to 4 or more adequate antidepressive treatments.
* The patient has a CGI severity of illness score of moderately ill (score of 4) or greater.
* The patient must be able to provide informed consent and complete all forms.

Exclusion Criteria:

* Patient has a history of schizophrenia, schizoaffective disorder, any other psychotic disorder, or a current major depressive episode that includes psychotic features; or is currently psychotic.
* Patient is currently enrolled in a double blind investigational study; patients who have completed the double-blind D-21 study will be allowed to enter the Registry for Long Term Follow-up
* Other than those patients who were enrolled in the D-21 study, patient has previously received VNS therapy.
* Patient has a history of rapid cycling bipolar disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic depression that is at least two years in duration or a recurrent depression that includes at least three lifetime episodes including the current major depressive episode (MDE); and an inadequate response to four or more adequate antidepressant treatments.
Sampling Method: Non-Probability Sample
Enrollment: 795 (Actual)
Dates: Start 2006-01; Primary Completion 2015-03 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam K. Ashton, MD, Principal Investigator — Suburban Psychiatric Associates; Herbert Ward, MD, Principal Investigator — University of Florida; Thomas Schwartz, MD, Principal Investigator — SUNY UMU at Syracuse; Mark Zetin, MD, Principal Investigator — Private Practice; Darin D. Dougherty, MD, Principal Investigator — Massachusetts General Hospital; George Keepers, MD, Principal Investigator — Oregon Health and Science University; Mustafa M. Husain, MD, Principal Investigator — UT Southwestern Medical Center at Dallas; Leighton Y. Huey, MD, Principal Investigator — UConn Health; James Kimball, MD, Principal Investigator — Wake Forest University Health Sciences; Peter J. Holland, MD, Principal Investigator — Florida Atlantic University; Robert Howland, MD, Principal Investigator — Western Psychiatric Institute & Clinic (WPIC); Anthony Rothschild, MD, Principal Investigator — University of Massachusetts, Worcester; Craig J Vine, MD, Principal Investigator — Psychiatric Recovery; Joel Young, MD, Principal Investigator — Rochester Center for Behavioral Science; Lawrence W Adler, MD, Principal Investigator — Clinical Insights; Harold Harsch, MD, Principal Investigator — Medical College of Wisconsin; Syed Ali, MD, Principal Investigator — Dupage Mental Health Services; Keming Gao, MD, Principal Investigator — University Hospitals Cleveland Medical Center; Todd M. Antin, M.D., DFAPA, Principal Investigator — Pact Atlanta, LLC; Basanti Basu, M.D., Principal Investigator — Century Health; Dwight Bearden, MD, Principal Investigator — Private Practice; David L. Dunner, MD, Principal Investigator — Center for Anxiety and Depression; Azfar Malik, MD, Principal Investigator — Psych Care Consultants Research; Joel Morgan, MD, Principal Investigator — Valdosta Psychiatric Associates LLC; Mark George, MD, Principal Investigator — Medical University of South Carolina; Frederick W. Reimherr, MD, Principal Investigator — Psychiatric & Behavorial Solutions; John Zajecka, MD, Principal Investigator — Psychiatric Medicine Associates, LLC; Michael Banov, MD, Principal Investigator — Northwest Behavioral Research Center; Robert Lehman, MD, Principal Investigator — Pharmasite Research, Inc.; Scott Aaronson, MD, Principal Investigator — Sheppard Pratt Health Systems, Inc.; Jaishree Narayanan, MD, Principal Investigator — Endeavor Health; Greg Seal, MD, Principal Investigator — Louisiana Clinical Research, LLC; Horacio Capote, MD, Principal Investigator — Dent Neurologic Institute; Charles Conway, MD, Principal Investigator — Washington University School of Medicine; Michael Lesem, MD, Principal Investigator — Claghorn-Lesem Reserach Clinic, Ltd.; Miguel Martelli, MD, Principal Investigator — MG Martelli, MD, PC and Associates; Ananda Pandurangi, MD, Principal Investigator — Virginia Commonwealth University; Peter Thompson, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio; Theodore Goodman, MD, Principal Investigator — Sutter Institute for Medical Research; Francisco Moreno, MD, Principal Investigator — University of Arizona; Martha Edelman, MD, Principal Investigator — Jamaica Hospital Medical Center; Peter Bulow, MD, Principal Investigator — Columbia University; Mark Bunker, Study Director — Cyberonics, Inc.; Mahendra Bhati, MD, Principal Investigator — University of Pennsylvania; Ronald Warnell, MD, Principal Investigator — Loma Linda University; Robert Cohen, MD, Principal Investigator — Cedars-Sinai Hospital; Janak Mehtani, MD, Principal Investigator — Fair Oaks Psychiatric Associates; Mounir Soliman, MD, Principal Investigator — University of California, San Diego; Francisco Fernandez, MD, Principal Investigator — University of South Florida; Arthur Holt, MD, Principal Investigator — Arthur Holt, Private Practice; Harold McGrath, MD, Principal Investigator — McGarth Clinic; Anthony D'Agostino, MD, Principal Investigator — Alexian Brothers Behavioral Health Hospital; Anne Gilbert, MD, Principal Investigator — 3c Methodist Hospital; Michael Burke, MD, Principal Investigator — Clinical Research Institute; Ed Coffey, MD, Principal Investigator — Henry Ford Health Services; Joseph Kwentus, MD, Principal Investigator — University of Mississippi Medical Center; David Ginsberg, MD, Principal Investigator — New York University of Medical Center; Melissa Martinez, MD, Principal Investigator — Baylor College of Medicine; Arnold Mech, MD, Principal Investigator — The Mech Center; Joseph Simpson, MD, Principal Investigator — Alamo Superior Research
Locations (55):
- United States (55):
  - University of Arizona, Tucson, Arizona
  - Cedars-Sinai Hospital, Beverly Hills, California
  - Mark Zetin, MD - Private Practice, Garden Grove, California
  - Loma Linda University, Loma Linda, California
  - Sutter Institute for Medical Research, Sacramento, California
  - Fair Oaks Psychiatric Associates, Sacramento, California
  - University of Connecticut Health Center, Farmington, Connecticut
  - Florida Atlantic University, Boca Raton, Florida
  - University of Florida, Gainesville, Florida
  - MG Martelli, MD, PC and Associates, Brunswick, Georgia
  - Arthur Holt, Private Practice, Columbus, Georgia
  - Pact Atlanta, LLC, Decatur, Georgia
  - Private Practice, Macon, Georgia
  - Northwest Behavioral Research Center, Marietta, Georgia
  - Valdosta Psychiatric Associates LLC, Valdosta, Georgia
  - Northshore University Health System, Evanston, Illinois
  - McGrath Clinic, Evergreen Park, Illinois
  - Alexian Brothers Behavioral Health Hospital, Hoffman Estates, Illinois
  - Psychiatric Medicine Associates, LLC, Skokie, Illinois
  - Dupage Mental Health Services, Wheaton, Illinois
  - 3c Methodist Hospital, Indianapolis, Indiana
  - Clinical Research Institute, Wichita, Kansas
  - Louisiana Clinical Research, LLC, Shreveport, Louisiana
  - Pharmasite Research Inc., Baltimore, Maryland
  - Sheppard Pratt Health Systems, Inc., Baltimore, Maryland
  - Clinical Insights, Glen Burnie, Maryland
  - Massachusetts General Hospital, Charlestown, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Rochester Center for Behavioral Medicine, Rochester Hills, Michigan
  - Psychiatric Recovery, Saint Paul, Minnesota
  - Precise Research Centers, Flowood, Mississippi
  - Washington University in St. Louis, St Louis, Missouri
  - Psych Care Consultants Research, St Louis, Missouri
  - Dent Neurologic Institute, Amherst, New York
  - Suburban Psychiatric Associates, Amherst, New York
  - Jamaica Hospital Medical Center, Jamaica, New York
  - Columbia University, New York, New York
  - SUNY UMU at Syracuse, Syracuse, New York
  - Wake Forest University - Health Sciences, Winston-Salem, North Carolina
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Century Health, Findlay, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Western Psychiatric Institute & Clinic (WPIC), Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - UT Southwestern Medical Center at Dallas, Dallas, Texas
  - Claghorn-Lesem Reserach Clinic, Ltd., Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - The Mech Center, Plano, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Alamo Superior Research, San Antonio, Texas
  - Psychiatric & Behavioral Solutions, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - Center for Anxiety and Depression, Mercer Island, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Background] Rush AJ, Sackeim HA, Marangell LB, George MS, Brannan SK, Davis SM, Lavori P, Howland R, Kling MA, Rittberg B, Carpenter L, Ninan P, Moreno F, Schwartz T, Conway C, Burke M, Barry JJ. Effects of 12 months of vagus nerve stimulation in treatment-resistant depression: a naturalistic study. Biol Psychiatry. 2005 Sep 1;58(5):355-63. doi: 10.1016/j.biopsych.2005.05.024. PMID 16139581
- [Background] Rush AJ, Marangell LB, Sackeim HA, George MS, Brannan SK, Davis SM, Howland R, Kling MA, Rittberg BR, Burke WJ, Rapaport MH, Zajecka J, Nierenberg AA, Husain MM, Ginsberg D, Cooke RG. Vagus nerve stimulation for treatment-resistant depression: a randomized, controlled acute phase trial. Biol Psychiatry. 2005 Sep 1;58(5):347-54. doi: 10.1016/j.biopsych.2005.05.025. PMID 16139580
- [Background] George MS, Rush AJ, Marangell LB, Sackeim HA, Brannan SK, Davis SM, Howland R, Kling MA, Moreno F, Rittberg B, Dunner D, Schwartz T, Carpenter L, Burke M, Ninan P, Goodnick P. A one-year comparison of vagus nerve stimulation with treatment as usual for treatment-resistant depression. Biol Psychiatry. 2005 Sep 1;58(5):364-73. doi: 10.1016/j.biopsych.2005.07.028. PMID 16139582
- [Background] Bajbouj M, Merkl A, Schlaepfer TE, Frick C, Zobel A, Maier W, O'Keane V, Corcoran C, Adolfsson R, Trimble M, Rau H, Hoff HJ, Padberg F, Muller-Siecheneder F, Audenaert K, van den Abbeele D, Matthews K, Christmas D, Eljamel S, Heuser I. Two-year outcome of vagus nerve stimulation in treatment-resistant depression. J Clin Psychopharmacol. 2010 Jun;30(3):273-81. doi: 10.1097/JCP.0b013e3181db8831. PMID 20473062
- [Derived] McAllister-Williams RH, Sousa S, Kumar A, Greco T, Bunker MT, Aaronson ST, Conway CR, Rush AJ. The effects of vagus nerve stimulation on the course and outcomes of patients with bipolar disorder in a treatment-resistant depressive episode: a 5-year prospective registry. Int J Bipolar Disord. 2020 May 2;8(1):13. doi: 10.1186/s40345-020-0178-4. PMID 32358769
- [Derived] Aaronson ST, Sears P, Ruvuna F, Bunker M, Conway CR, Dougherty DD, Reimherr FW, Schwartz TL, Zajecka JM. A 5-Year Observational Study of Patients With Treatment-Resistant Depression Treated With Vagus Nerve Stimulation or Treatment as Usual: Comparison of Response, Remission, and Suicidality. Am J Psychiatry. 2017 Jul 1;174(7):640-648. doi: 10.1176/appi.ajp.2017.16010034. Epub 2017 Mar 31. PMID 28359201

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The TRD Registry was to enroll over a maximum period of 6 years & patients were to be followed for at least 60 months. All sites were to first recruit patients who had agreed to have adjunctive VNS Therapy. Sites were also asked to enroll patients with TRD who would not be implanted with VNS Therapy and would act as a concurrent control group.
Pre-assignment Details: A total of 878 subjects were screened in the TRD Registry Study. Thirty-seven were not eligible and 46 were eligible but not treated for various reasons. This left a total of 795 patients in the Safety Population (SP).
Groups:
- VNS Therapy: Disposition of study patients from baseline to the end of the study. The VNS Therapy arm, was comprised of D-23 Original patients (Patients that entered the TRD Registry without previous VNS Therapy treatment and selected the VNS Therapy study arm) and D-21 Rollover patients (Patients that entered the TRD Registry, having previously participated in the D-21 study-NCT00305565 and still being treated with VNS Therapy).
- Treatment as Usual (TAU): Disposition of study patients from baseline to the end of the study. The TAU arm were subjects that entered the TRD Registry without previous VNS Therapy treatment and selected the TAU study arm.
Period: Overall Study
Arm/Group | VNS Therapy | Treatment as Usual (TAU)
Started | 494 | 301
VNS Therapy D-23 Original | 335 | 0
VNS Therapy D-21 (NCT00305565) Rollovers | 159 | 0
Completed | 299 | 138
Not Completed | 195 | 163
Not completed — Physician Decision | 4 | 7
Not completed — Death | 7 | 8
Not completed — Withdrawal by Subject | 55 | 37
Not completed — Non-Compliance | 40 | 39
Not completed — Did not Meet (I/E) | 3 | 1
Not completed — Other (i.e. lost to f/u, site closure) | 86 | 71

BASELINE CHARACTERISTICS:
Population: A total of 878 subjects were screened. Thirty-seven were not eligible and 46 were eligible but not treated for various reasons. This left a total of 795 patients in the Safety Population (SP). The total number of patients in each group may be lower than SP if there was missing D-21 assessment data, as D-21 baseline data was not identical to D-23.
Groups:
- VNS Therapy D-23 Original: Subjects that entered the TRD Registry without previous VNS Therapy treatment and selected the VNS Therapy study arm.
- VNS Therapy D-21 Rollover: Subjects that entered the TRD Registry, having previously participated in the D-21 study and still being treated with VNS Therapy treatment were included within the VNS Therapy group. Based on the duration from initial implant to enrollment date, the D-21 rollover patients entered at the appropriate D-23 follow-up interval (i.e., patient enrolls at 24 months post implant for their first D-23 follow up visit. This 24 month visit corresponds to the 24 month follow up in the TRD Registry). Starting with the first TRD Registry visit, the D-21 long-term patients were to follow the same data collection schedule as other Original VNS and TAU Registry patients.
- Treatment as Usual (TAU): Non-VNS Patients - Treatment-resistant depression patients not receiving VNS Therapy. Subjects that entered the TRD Registry without previous VNS Therapy treatment and selected the TAU study arm.
- Total: Total of all reporting groups
Arm/Group | VNS Therapy D-23 Original | VNS Therapy D-21 Rollover | Treatment as Usual (TAU) | Total
Number analyzed (Participants) | 335 | 159 | 301 | 795
Age, Customized [Mean (Standard Deviation); unit: Years]
  Age at Baseline (n=335, n=159, n=301) | 48.9 (10.41) | 48.9 (9.51) | 49.9 (11.07) | 49.3 (10.49)
  Age-Initial Onset of Depression(n=334,n=159,n=301) | 20.8 (12.13) | 21.1 (11.11) | 21.1 (11.40) | 21.0 (11.64)
  Age-Initial Dx. of Depression(n=334,n=159,n=301) | 29.0 (10.95) | 28.6 (10.50) | 29.5 (11.89) | 29.1 (11.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 231 | 119 | 211 | 561
  Male | 104 | 40 | 90 | 234
Race/Ethnicity, Customized [Number; unit: Participants] — Ethnic Orgin of participants in the study
  Participants
    Caucasian | 323 | 155 | 274 | 752
    African-American | 4 | 4 | 6 | 14
    Hispanic | 3 | 0 | 19 | 22
    Asian | 2 | 0 | 1 | 3
    Other | 3 | 0 | 1 | 4
Lifetime Episodes of Depression Diagnosed (n=335, n=0, n=301) [Mean (Standard Deviation); unit: Lifetime Episodes of Depression] | 14.9 (24.14) | NA (NA) — This Variable was captured as categorical variable as part of D-21 study | 12.0 (23.86) | 13.5 (24.03)
Number of Failed Treatments (n=335, n=159, n=301) [Mean (Standard Deviation); unit: Number of Failed Treatments] | 8.0 (3.05) | 8.6 (3.74) | 7.3 (2.92) | 7.9 (3.19)
Suicide Attempts in Lifetime (n=335, n=159, n=301) [Mean (Standard Deviation); unit: Number of Suicide Attempts in a Lifetime] | 2.1 (4.38) | 1.2 (2.95) | 1.2 (2.41) | 1.6 (3.49)
Diagnosis Disorder (Major Depressive Disorder (MDD) or Bipolar Disorder (BPD) [Number; unit: Participants]
  MDD, Recurrent, Moderate Severity | 42 | 21 | 69 | 132
  MDD, Recurrent, Severe w/o Psychotic Features | 135 | 90 | 95 | 320
  MDD, Single Episode, Moderate Severity | 12 | 4 | 30 | 46
  MDD, Single Episode, Severe w/o Psychotic Features | 49 | 7 | 36 | 92
  BPD I, MRE Depressed, Moderate Severity | 19 | 6 | 21 | 46
  BPD I, MRE Depressed,Severe w/o Psychotic Features | 46 | 16 | 12 | 74
  BPD II, MRE Depressed | 32 | 15 | 38 | 85

OUTCOME MEASURES:

1. Primary Outcome: Montgomery Asberg Depression Rating Scale (MADRS)% Responders (>/= 50% Improvement From Baseline)
Description: Response Rate was computed and summarized as the proportion of patients that achieved ≥ 50% reduction from baseline in MADRS total score at each post-baseline visit. The MADRS is a ten-item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders. Higher MADRS score indicates more severe depression, and each item yields a score of 0 to 6. The overall score ranges from 0 to 60. The lower a score the less symptom severity is seen. A patient was considered a "Responder" (Yes = 1) if achieved ≥ 50% reduction from baseline in MADRS total score at visit month assessment post-baseline. A "Non-Responder" (No = 0) was any patient who did not achieve ≥ 50% reduction from baseline in MADRS score at visit month assessment post-baseline.
  Total number of patients in each group may be lower than ITT in a case of missing assessment data.
Time Frame: 3-Month Through 60-Month (Post Baseline)
Population: Intent-To-Treat (ITT) Population: VNS Therapy Population (n=489 (D-23=330 + D-21=159)) + (n= 276) TAU population
Measure: Number; unit: Percentage of Participants
Groups:
- VNS Therapy; Treatment As Usual (TAU): MADRS % Responders (Percentage of Responders)
Arm/Group | VNS Therapy | Treatment As Usual (TAU)
Number analyzed (Participants) | 489 | 276
Percentage of Participants
  3-Month (n=454, n=249) | 24 | 8.8
  6-Month (n=432, n=224) | 28 | 13.8
  9-Month (n=408, n=193) | 33.8 | 13.5
  12-Month (n=403, n=194) | 38.2 | 17.5
  18-Month (n=223, n=162) | 34.1 | 15.4
  24-Month (n=233, n=146) | 38.6 | 18.5
  30-Month (n=224, n=138) | 34.8 | 22.5
  36-Month (n=245, n=133) | 38.8 | 17.3
  42-Month (n=245, n=121) | 41.2 | 19.0
  48-Month (n=246, n=109) | 46.3 | 22.0
  54-Month (n=222, n=102) | 48.2 | 27.5
  60-Month (n=250, n=116) | 49.6 | 25.9
Statistical Analysis 1: Comparison: VNS Therapy; Null Hypothesis: Percentage of responders across groups is the same. Alternate Hypothesis: Percentage of responders across groups is different; Test type: Superiority or Other; MMRM Least Squares Mean = 38.1, 95% CI 2-sided [36.3 to 39.9] — Mixed Model Repeated Measure analysis on MADRS responders (binary variable with 1=yes, 0=no) as the response variable in the model. The covariates are treatment, visit and propensity quintile. This analysis of covariance produced least square means
Statistical Analysis 2: Comparison: Treatment As Usual (TAU); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; MMRM Least Squares Mean = 17.0, 95% CI 2-sided [15.2 to 19.0] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: VNS Therapy vs Treatment As Usual (TAU); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < .0001, ANCOVA

2. Secondary Outcome: Time Until Recurrence (TUR) for Patients That Achieved Remission, Based on Montgomery Asberg Depression Rating Scale (MADRS)
Description: Recurrence based on MADRS is defined as first time attained MADRS total score ≥ 20 after achieving remission. Remission is a binary outcome response variable (Yes/No in-remission) defined as MADRS total score </= 9 at visit month assessment post-baseline. Duration of remission Computed as recorded date of the first recurrence/relapse (MADRS score >/= 20) minus the recorded date of first achieved remission (MADRS score </=9). Only a subpopulation that achieved remission will be included in the summary.
  Time-to-event analyses were summarized using Kaplan-Meier curves. Patients who did not achieve recurrence at the end of the study were censored on the last visit date recorded. Additionally, patients who discontinued early were censored on last date of contact. Censored observations and confidence intervals for the estimated median times were calculated.
Time Frame: 3-Month Through 60-Month (Post Baseline)
Population: Intent-To-Treat (ITT) Population: VNS Therapy Population (n=489 (D-23=330 + D-21=159)) + (n= 276) TAU population
Measure: Median (95% Confidence Interval); unit: Months
Units Other Than Participants: Censored Patients
Groups:
- VNS Therapy; Treatment As Usual (TAU): Time until recurrence based on the MADRS
Arm/Group | VNS Therapy | Treatment As Usual (TAU)
Number analyzed (Participants) | 204 | 70
Number analyzed (Censored Patients) | 151 | 46
Months
  1st Quartile (25%);Time (Mo.) Until Recurrence | 14 [10 to 19] | 9 [6 to 13]
  Kaplan-Meier Median;Time (Mo.) Until Recurrence | 40 [26 to NA] — Unable to compute based on Kaplan Meier Calculation due to too few events | 19 [10 to NA] — Unable to compute based on Kaplan Meier Calculation due to too few events.
Statistical Analysis 1: Comparison: VNS Therapy vs Treatment As Usual (TAU); Test type: Superiority or Other; p = 0.1015, Log Rank — Comparison for Kaplan Meier Median Time until recurrence; Null hypothesis: median TUR between 2 groups is not different. Alternate hypothesis: median TUR between 2 groups is different

3. Secondary Outcome: Montgomery Asberg Depression Rating Scale (MADRS)% Remitters (MADRS Total Score ≤9 at Visit Month Assessment Post-Baseline)
Description: Remission is a binary outcome response variable (Yes/No Inremission) defined as MADRS total score < 9 at visit month assessment post-baseline. The MADRS is a ten-item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders. Higher MADRS score indicates more severe depression, and each item yields a score of 0 to 6. The overall score ranges from 0 to 60. The lower a score the less symptom severity is seen and in general it is accepted that a score between 0-6 is indicative of a normal/symptom-free individual; 7-19 is indicative of a patient with mild depression; 20-34 is indicative of a patient with moderate depression; and >34 is indicative of a patient with severe depression. Total number of patients in each group may be lower than ITT in a case of missing assessment data.
Time Frame: 3-Month Through 60-Month (Post Baseline)
Population: Intent-To-Treat (ITT) Population: VNS Therapy Population (n=489 (D-23=330 + D-21=159)) + (n= 276) TAU population
Measure: Number; unit: Percentage of Participants
Groups:
- VNS Therapy; Treatment As Usual (TAU): MADRS % Remitters (Percentage of Subjects in Remission)
Arm/Group | VNS Therapy | Treatment As Usual (TAU)
Number analyzed (Participants) | 489 | 276
Percentage of Participants
  3-Month (n=454, n=249) | 8.6 | 2.8
  6-Month (n=432, n=224) | 15 | 6.3
  9-Month (n=408, n=193) | 16.2 | 5.7
  12-Month (n=403, n=194) | 19.4 | 8.2
  18-Month (n=223, n=162) | 14.3 | 7.4
  24-Month (n=233, n=146) | 21.9 | 11
  30-Month (n=224, n=138) | 20.5 | 12.3
  36-Month (n=245, n=133) | 19.2 | 11.3
  42-Month (n=245, n=121) | 24.9 | 13.2
  48-Month (n=246, n=109) | 25.6 | 14.7
  54-Month (n=222, n=102) | 28.4 | 13.7
  60-Month (n=250, n=116) | 27.6 | 19
Statistical Analysis 1: Comparison: VNS Therapy; Null Hypothesis: Percentage of remitters across groups is the same. Alternate Hypothesis: Percentage of remitters across groups is different; Test type: Superiority or Other; MMRM Least Squares Mean = 19.8, 95% CI 2-sided [18.4 to 21.3] — Mixed Model Repeated Measure analysis on MADRS remitters (binary variable with 1=yes, 0=no) as the response variable in the model. The covariates are treatment, visit and propensity quintile. This analysis of covariance produced least square means
Statistical Analysis 2: Comparison: Treatment As Usual (TAU); [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; MMRM Least Squares Mean = 8.1, 95% CI 2-sided [6.9 to 9.5] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: VNS Therapy vs Treatment As Usual (TAU); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < .0001, ANCOVA

4. Post Hoc Outcome: Mortality and Suicidality in Safety Population (Total Number of Deaths)
Description: The number of deaths on the study were collected from the baseline visit.
Time Frame: 3-Month (baseline or implantation) Through 60-Month (Post Baseline)
Population: Safety Population (SP): VNS Therapy Population (n=494 (D-23=335 + D-21=159)) + (n= 301) TAU population
Measure: Number; unit: Number of Deaths
Groups:
- VNS Therapy: VNS Patients - Treatment-resistant depression patients treated with VNS Therapy
- Treatment as Usual (TAU): Non-VNS Patients - Treatment-resistant depression patients not receiving VNS Therapy
Arm/Group | VNS Therapy | Treatment as Usual (TAU)
Number analyzed (Participants) | 494 | 301
Number of Deaths | 7 | 8

5. Post Hoc Outcome: Mortality and Suicidality in Safety Population (Total Patient Years Exposed)
Description: Treatment exposure time in years for all patients for all treatment groups were calculated in 1000 person year measure.
Time Frame: 3-Month Through 60-Month (Post Baseline)
Population: Safety Population (SP): VNS Therapy Population (n=494 (D-23=335 + D-21=159)) + (n= 301) TAU population
Measure: Number; unit: Exposure Per 1000 Patient Years
Arm/Group | VNS Therapy | Treatment as Usual (TAU)
Number analyzed (Participants) | 494 | 301
Exposure Per 1000 Patient Years | 1985.083 | 926.493

6. Post Hoc Outcome: Mortality and Suicidality in Safety Population (All-Cause Mortality/1000 Person Years)
Description: All cause mortality is defined as the number of deaths per calculated 1000 person years.
Time Frame: 3-Month Through 60-Month (Post Baseline)
Population: Safety Population (SP): VNS Therapy Population (n=494 (D-23=335 + D-21=159)) + (n= 301) TAU population
Measure: Number; unit: Deaths Per 1000 Person Years
Arm/Group | VNS Therapy | Treatment as Usual (TAU)
Number analyzed (Participants) | 494 | 301
Deaths Per 1000 Person Years | 3.53 | 8.63

7. Post Hoc Outcome: Mortality and Suicidality in Safety Population (Number of Suicides)
Description: The number suicides on the study were collected from the baseline visit.
Time Frame: 3-Month Through 60-Month (Post Baseline)
Population: Safety Population (SP): VNS Therapy Population (n=494 (D-23=335 + D-21=159)) + (n= 301) TAU population
Measure: Number; unit: Number of Suicides
Arm/Group | VNS Therapy | Treatment as Usual (TAU)
Number analyzed (Participants) | 494 | 301
Number of Suicides | 2 | 2

8. Post Hoc Outcome: Mortality and Suicidality in Safety Population (Suicides/1000 Person Years)
Description: The number of suicides per calculated 1000 person years.
Time Frame: 3-Month Through 60-Month (Post Baseline)
Population: Safety Population (SP): VNS Therapy Population (n=494 (D-23=335 + D-21=159)) + (n= 301) TAU population
Measure: Number; unit: Number of Suicides Per 1000 Person Years
Arm/Group | VNS Therapy | Treatment as Usual (TAU)
Number analyzed (Participants) | 494 | 301
Number of Suicides Per 1000 Person Years | 1.01 | 2.20

9. Secondary Outcome: Predictors of Suicidality Based on Montgomery Asberg Depression Rating Scale (MADRS) Item 10 Score - Baseline MADRS Item 10 Suicidal Ideation
Description: This assessment was completed telephonically by a third party rater (Central Rater Group). The rating was based on a clinical interview moving from broadly phrased questions about symptoms to more detailed ones, which allowed a precise rating of severity. The rater decided whether the rating lied on the defined scale steps (0, 2, 4, 6) or between them (1, 3, 5) and then checked the appropriate selection on the MADRS Item 10 Suicidal Thoughts (Ideation).
  Total number of patients analyzed may be lower than ITT in a case of missing assessment data.
Time Frame: 1 Week Pre-Baseline
Population: D-23 Original + TAU [(n= 330) + (n= 276)] minus 2 missing assessment data. These risk factors assessed at baseline and pre-baseline were not collected with respect to treatment, therefore this information is not presented by treatment arm.
Measure: Number; unit: Percentage of Patients
Groups:
- ITT Population: VNS Therapy and Treatment as Usual (TAU)
Arm/Group | ITT Population
Number analyzed (Participants) | 763
Percentage of Patients
  0 Enjoys Life | 6.03
  1 | 28.83
  2 Weary of Life | 25.56
  3 | 18.87
  4 Probably Better Off Dead | 14.81
  5 | 4.72
  6 Explicit Plans for Suicide | 1.18
Statistical Analysis 1: Comparison: ITT Population; The statistical modeling of predictors of suicide attempts and suicidal ideations considered 15 variables, defined in the protocol a priori to determine which ones were predictive of suicide attempts and suicidal ideations. Four variables representing the baseline disease and patient factors were considered predictors of suicidality. This outcome measure presents the underlying data collected and the corresponding correlation coefficient for one of the 4 variables identified; Test type: Superiority or Other; p < 0.0001, Pearson Correlation Coefficients — Null hypothesis: There is a correlation between MADRS follow-up suicidal thoughts and baseline suicidal thoughts. Alternate hypothesis: There is no correlation between MADRS follow-up suicidal thoughts and baseline suicidal thoughts; Pearson Correlation Coefficients = .34997

10. Post Hoc Outcome: Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF) Change From Baseline by Visit Month
Description: The Q-LES-Q-SF is a self-report scale to assess the degree of enjoyment and satisfaction experienced by the patient during the past week. There are 2 forms of this instrument: the short form and the long form. The short form employs the 14 general activities included in the long form, as well as 2 global items. Five-point item scores (1 to 5) are aggregated, with higher scores indicative of greater enjoyment or satisfaction in each domain. The scoring of the Q-LESQ-SF involves summing only the first 14 items to yield a raw total score. The last 2 items are not included in the total score but stand alone. The raw total score ranges from 14 (worst score) to 70 (best score). Higher Q-LES-QSF score indicates more enjoyment and satisfaction (Endicott, Nee et al. 1993).
Time Frame: 3-Month Through 60-Month (Post Baseline)
Population: ITT Population minus D-21 Subjects: VNS Therapy Population (D-23=330) + (n= 276) TAU population. The total number of patients in each group is lower than ITT due to missing assessment data, for which a large portion is that of D-21 subjects. The Q-LES-Q-SF was not collected in the D-21 Study.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- VNS Therapy; Treatment As Usual (TAU): Change from Baseline Score
Arm/Group | VNS Therapy | Treatment As Usual (TAU)
Number analyzed (Participants) | 330 | 276
units on a scale
  3 Months (n=322, n=261) | 7.92 (16.20) | 1.38 (16.61)
  6 Months (n=298, n=239) | 9.11 (15.66) | 4.36 (17.46)
  9 Months (n=270, n=216) | 10.50 (16.74) | 3.97 (17.07)
  12 Months (n=266, n=211) | 11.04 (18.36) | 5.49 (17.56)
  18 Months (n=264, n=179) | 11.40 (18.29) | 3.88 (16.03)
  24 Months (n=240, n=159) | 13.15 (18.13) | 7.50 (16.73)
  30 Months (n=223, n=147) | 13.06 (18.63) | 8.13 (16.73)
  36 Months (n=219, n=149) | 15.59 (18.43) | 8.34 (16.11)
  42 Months (n=196, n=141) | 14.67 (17.46) | 8.55 (17.95)
  48 Months (n=179, n=127) | 14.70 (19.02) | 9.88 (17.28)
  54 Months (n=156, n=128) | 16.44 (18.63) | 10.49 (16.74)
  60 Months (n=173, n=136) | 17.20 (17.59) | 10.11 (17.93)
Statistical Analysis 1: Comparison: VNS Therapy vs Treatment As Usual (TAU); 3 Month Time point; Test type: Superiority or Other; p < .0001, F-Test — Null Hypothesis: Difference between change from baseline value of two treatment groups equals zero. Alternate Hypothesis: Difference between change from baseline value of two treatment groups is not equal to zero
Statistical Analysis 2: Comparison: VNS Therapy vs Treatment As Usual (TAU); 6 Month Time point; Test type: Superiority or Other; p = .0068, F-Test — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: VNS Therapy vs Treatment As Usual (TAU); 9 Month Time point; Test type: Superiority or Other; p = .0008, F-Test — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 4: Comparison: VNS Therapy vs Treatment As Usual (TAU); 12 Month Time point; Test type: Superiority or Other; p = .0003, F-Test — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 5: Comparison: VNS Therapy vs Treatment As Usual (TAU); 18 Month Time point; Test type: Superiority or Other; p < .0001, F-Test — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 6: Comparison: VNS Therapy vs Treatment As Usual (TAU); 24 Month Time point; Test type: Superiority or Other; p = .0059, F-Test — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 7: Comparison: VNS Therapy vs Treatment As Usual (TAU); 30 Month Time point; Test type: Superiority or Other; p = .0028, F-Test — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 8: Comparison: VNS Therapy vs Treatment As Usual (TAU); 36 Month Time point; Test type: Superiority or Other; p = .0002, F-Test — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 9: Comparison: VNS Therapy vs Treatment As Usual (TAU); 42 Month Time point; Test type: Superiority or Other; p = .0051, F-Test — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 10: Comparison: VNS Therapy vs Treatment As Usual (TAU); 48 Month Time point; Test type: Superiority or Other; p = .0363, F-Test — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 11: Comparison: VNS Therapy vs Treatment As Usual (TAU); 54 Month Time point; Test type: Superiority or Other; p = .0048, F-Test — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 12: Comparison: VNS Therapy vs Treatment As Usual (TAU); 60 Month Time point; Test type: Superiority or Other; p = .0009, F-Test — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 13: Comparison: VNS Therapy; Null Hypothesis: Difference between change from baseline value of two treatment groups equals zero. Alternate Hypothesis: Difference between change from baseline value of two treatment groups is not equal to zero; Test type: Superiority or Other; MMRM Least Squares Mean = 12.1009, 95% CI 2-sided [10.8979 to 13.3039] — Mixed Model Repeated Measure analysis on Q-LES-Q change from baseline score (continuous var) as the response variable in the model. The covariates are treatment, visit and propensity quintile. This analysis of covariance produced least square means
Statistical Analysis 14: Comparison: Treatment As Usual (TAU); [analysis description as in outcome 10, analysis 13]; Test type: Superiority or Other; MMRM Least Squares Mean = 7.5964, 95% CI 2-sided [6.1327 to 9.0602] — [estimate comment as in outcome 10, analysis 13]
Statistical Analysis 15: Comparison: VNS Therapy vs Treatment As Usual (TAU); [analysis description as in outcome 10, analysis 13]; Test type: Superiority or Other; p < .0001, ANCOVA

11. Secondary Outcome: Predictors of Suicidality Based on Montgomery Asberg Depression Rating Scale (MADRS) Item 10 Score - Medical Threat to Life of Most Recent Suicidal Gesture
Description: This assessment was completed by the physician at the baseline visit in a clinical interview. The physician decided which category (as shown in outcome measure data table) best characterized the patient's medical threat to life of their most recent suicidal gesture or attempt.
  Total number of patients analyzed may be lower than ITT in a case of missing assessment data.
Time Frame: Baseline
Population: D-23 Original + TAU [(n= 330) + (n= 276)] minus 159 missing assessment data. These risk factors assessed at baseline and pre-baseline were not collected with respect to treatment, therefore this information is not presented by treatment arm.
Measure: Number; unit: Percentage of Patients
Arm/Group | ITT Population
Number analyzed (Participants) | 606
Percentage of Patients
  Patient Never Made an Attempt | 46.70
  No Information or Not Sure | 3.14
  No Danger | 5.61
  Minimal | 3.47
  Mild | 8.91
  Moderate | 18.15
  Severe | 11.39
  Extreme | 2.64
Statistical Analysis 1: Comparison: ITT Population; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p < .0001, Pearson Correlation Coefficients — Null hypothesis: There is a correlation between MADRS follow-up suicidal thoughts and baseline medical threat to life. Alternate hypothesis: There is no correlation between MADRS follow-up suicidal thoughts and baseline medical threat to life; Pearson Correlation Coefficients = .14837

12. Secondary Outcome: Predictors of Suicidality Based on Montgomery Asberg Depression Rating Scale (MADRS) Item 10 Score - Intent of Most Recent Suicidal Gesture
Description: This assessment was completed by the physician at the baseline visit in a clinical interview. The physician decided which category (as shown in outcome measure data table) best characterized the patient's intent of their most recent suicidal gesture or attempt.
  Total number of patients analyzed may be lower than ITT in a case of missing assessment data.
Time Frame: Baseline
Population: as for outcome 11
Measure: Number; unit: Percentage of Patients
Arm/Group | ITT Population
Number analyzed (Participants) | 606
Percentage of Patients
  Patient Never Made an Attempt | 46.86
  No Information or Not Sure | 3.80
  Obviously no Intent | 2.31
  Not Sure or Only Minimal Intent | 5.12
  Definite But Very Ambivalent | 11.06
  Serious | 12.05
  Very Serious | 9.57
  Extreme | 9.24
Statistical Analysis 1: Comparison: ITT Population; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p < .0001, Pearson Correlation Coefficients — Null hypothesis: There is a correlation between MADRS f/u suicidal thoughts and baseline intent of suicidal gesture. Alternate hypothesis: There is no correlation between MADRS f/u suicidal thoughts and baseline intent of suicidal gesture; Pearson Correlation Coefficients = .14819

13. Secondary Outcome: Predictors of Suicidality Based on Montgomery Asberg Depression Rating Scale (MADRS) Item 10 Score - Primary Diagnosis of MDE
Description: This assessment was completed by the physician at the screening visit. The physician decided which DSM-IV Diagnosis (as shown in outcome measure data table) best characterized the patient's primary diagnosis of MDE.
Time Frame: Screening
Population: D-23 Original + TAU [(n= 330) + (n= 276)]. These risk factors assessed at baseline and pre-baseline were not collected with respect to treatment, therefore this information is not presented by treatment arm.
Measure: Number; unit: Percentage of Patients
Arm/Group | ITT Population
Number analyzed (Participants) | 765
Percentage of Patients
  MDD, Recurrent, Moderate Severity | 16.99
  MDD, Recurrent, Severe w/o Psychotic Features | 40.39
  MDD, Single Episode, Moderate Severity | 5.88
  MDD, Single Episode, Severe w/o Psychotic Features | 11.24
  BPD I, MRE Depressed, Moderate Severity | 5.75
  BPD I, MRE Depressed,Severe w/o Psychotic Features | 9.41
  BPD II, MRE Depressed | 10.33
Statistical Analysis 1: Comparison: ITT Population; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = .0012, Pearson Correlation Coefficients — Null hypothesis: There is a correlation between MADRS follow-up suicidal thoughts and baseline primary diagnosis of MDE. Alternate hypothesis: There is no correlation between MADRS follow-up suicidal thoughts and baseline primary diagnosis of MDE; Pearson Correlation Coefficients = .04625

ADVERSE EVENTS:
Time Frame: N/A (Adverse event information was not collected as part of the TRD Registry Protocol)
Description: Physicians were instructed to notify Cyberonics' Clinical Technical Support (CTS) department of all Medical Devices Reporting (MDR) events that occurred in TRD Registry participants receiving VNS Therapy.
Groups:
- Safety Events: N/A (not collected)
Arm/Group | Safety Events
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No